CLINICAL TRIAL: NCT04902989
Title: Association Between Environmental Pollutants and Their Effects on Respiratory
Brief Title: Environmental Pollutants and Their Effects on Respiratory Allergy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cindy Elizabeth de Lira-Quezada (Other)
Collaborators: Medicina (Other)
Responsible Party: Sponsor-Investigator, Cindy Elizabeth de Lira-Quezada, Professor of Allergy and Clinical Immunology, Medicina
Organization: Medicina (Other)
Other Study IDs: AL2100004
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Allergic Rhinitis; Allergic Asthma; Pollution; Exposure
Keywords: pollutants; allergy; symptoms
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity | interventions — Environmental Pollutants; Propolis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pollutants and pollen — Pollutants (ozone, SO3, NO3, PM2.5, diesel exhaust particles)

SUMMARY:
In Latin America and the Caribbean, more than 100 million people are exposed to higher levels of pollution than those recommended by WHO. The objective of the study is to determine the relationship between exposure to environmental pollutants and the prevalence and exacerbation of respiratory allergy. It is an observational, prospective, longitudinal and descriptive study that will include subjects older than 6 years who come to the consultation of the Regional Center for Allergy and Clinical Immunology with a diagnosis of respiratory allergy, positive skin tests and who live in Monterrey and its metropolitan area. After verbal assent, the subject's address and work area will be registered, the Rhinitis Control Assessment Test and the Asthma Control Test as well as spirometry will be made. The geolocation of industries and avenues near the address and work area of subjects will be carried out, as well as the determination of pollutants and pollens by the Integral Monitoring System (SIMA) and the Pollen Sense device. Subsequently, the correlation between exposure to pollutants and respiratory allergy will be analyzed. Dispersion models will be built considering pollutants and climatic factors (precipitation, wind speed, humidity and temperature). By carrying out this project, it will be possible to contribute to the identification of the factors that lead to the development and exacerbation of allergic respiratory diseases and subsequently propose the implementation of measures for their control and recommendations for prevention to the population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 6 years of age who attend the the Regional Center of Allergy and Clinical Immunology of the University Hospital "Dr. José Eleuterio González "with a diagnosis of respiratory allergy (allergic rhinitis and asthma) and type I immunological hypersensitivity demonstrated by skin tests by an allergist; and who live in the city of Monterrey and its metropolitan area.

Exclusion Criteria:

* Subjects for whom it is not possible to perform a pulmonary function test or who have concomitant diseases such as COPD, heart disease or some other pathology that, in the opinion of the investigator, may cause confusion with respiratory symptoms. Patients with negative skin tests to aeroallergens.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects older than 6 years of age, who attend the Regional Center of Allergy and Clinical Immunology of the University Hospital "Dr. José Eleuterio González "with a diagnosis of respiratory allergy (allergic rhinitis and asthma) and type I immunological hypersensitivity demonstrated by skin tests performed by an allergist and who live in Monterrey or its metropolitan area.
  They will be invited to participate in the protocol and if they agree to be included, they will respond to informed verbal consent or assent.
Sampling Method: Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-08-10 (Estimated); Study Completion 2022-08-10 (Estimated)

PRIMARY OUTCOMES:
Association of respiratory symptoms with exposure to pollutants and pollen | 1 year
  To determine the relationship between exposure to environmental pollutants and the prevalence and exacerbation of respiratory allergy.

SECONDARY OUTCOMES:
Avenues with highest diesel exhaust particles and traffic related particles | 1 year
  Locate the avenues with the highest flow and vehicular load releasing diesel removal particles (DEP) and traffic-related air pollutants (TRAP).
Location of the main industries that emit pollutants | 1 year
  Location of the main industries that emit pollutants of particulate matter (PM), nitrogen dioxide (NO2), sulfur dioxide (SO2), carbon monoxide (CO) and ozone (O3).
Distance of greater exposure to pollutants | 1 year
  To assess the relationship between the distance to PM, traffic-related air pollutants (TRAP) and diesel exhaust particles (DEP) with the prevalence of respiratory allergy symptoms with home and work address.
Time of pollutant exposure and association with respiratory symptoms | 1 year
  Evaluate the relationship between the time of exposure to PM, NO2, SO2, O3, traffic-related air pollutants (TRAP) and diesel exhaust particles (DEP) with the prevalence of respiratory allergy symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra N Gonzalez Diaz, MD,PhD, Study Director — Head of the Allergy and Clinical Immunology Service
Locations (1):
- Regional Center of Allergy and Clinical Immunology, Hospital Universitario "Dr. José Eleuterio González", Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cecchi L, D'Amato G, Annesi-Maesano I. External exposome and allergic respiratory and skin diseases. J Allergy Clin Immunol. 2018 Mar;141(3):846-857. doi: 10.1016/j.jaci.2018.01.016. PMID 29519451
- [Background] Lai CK, Beasley R, Crane J, Foliaki S, Shah J, Weiland S; International Study of Asthma and Allergies in Childhood Phase Three Study Group. Global variation in the prevalence and severity of asthma symptoms: phase three of the International Study of Asthma and Allergies in Childhood (ISAAC). Thorax. 2009 Jun;64(6):476-83. doi: 10.1136/thx.2008.106609. Epub 2009 Feb 22. PMID 19237391
- [Background] Traina G, Barbalace A, Betti F, Bolzacchini E, Bonini M, Contini D, Felice G, Foti T, Mantecca P. What impact of air pollution in pediatric respiratory allergic diseases. Pediatr Allergy Immunol. 2020 Nov;31 Suppl 26:26-28. doi: 10.1111/pai.13362. PMID 33236436
- [Background] D'Amato G, Bergmann KC, Cecchi L, Annesi-Maesano I, Sanduzzi A, Liccardi G, Vitale C, Stanziola A, D'Amato M. Climate change and air pollution: Effects on pollen allergy and other allergic respiratory diseases. Allergo J Int. 2014;23(1):17-23. doi: 10.1007/s40629-014-0003-7. Epub 2014 Feb 19. PMID 26120514
- [Background] Landrigan PJ, Fuller R, Acosta NJR, Adeyi O, Arnold R, Basu NN, Balde AB, Bertollini R, Bose-O'Reilly S, Boufford JI, Breysse PN, Chiles T, Mahidol C, Coll-Seck AM, Cropper ML, Fobil J, Fuster V, Greenstone M, Haines A, Hanrahan D, Hunter D, Khare M, Krupnick A, Lanphear B, Lohani B, Martin K, Mathiasen KV, McTeer MA, Murray CJL, Ndahimananjara JD, Perera F, Potocnik J, Preker AS, Ramesh J, Rockstrom J, Salinas C, Samson LD, Sandilya K, Sly PD, Smith KR, Steiner A, Stewart RB, Suk WA, van Schayck OCP, Yadama GN, Yumkella K, Zhong M. The Lancet Commission on pollution and health. Lancet. 2018 Feb 3;391(10119):462-512. doi: 10.1016/S0140-6736(17)32345-0. Epub 2017 Oct 19. No abstract available. PMID 29056410
- [Background] D'Amato G, Holgate ST, Pawankar R, Ledford DK, Cecchi L, Al-Ahmad M, Al-Enezi F, Al-Muhsen S, Ansotegui I, Baena-Cagnani CE, Baker DJ, Bayram H, Bergmann KC, Boulet LP, Buters JT, D'Amato M, Dorsano S, Douwes J, Finlay SE, Garrasi D, Gomez M, Haahtela T, Halwani R, Hassani Y, Mahboub B, Marks G, Michelozzi P, Montagni M, Nunes C, Oh JJ, Popov TA, Portnoy J, Ridolo E, Rosario N, Rottem M, Sanchez-Borges M, Sibanda E, Sienra-Monge JJ, Vitale C, Annesi-Maesano I. Meteorological conditions, climate change, new emerging factors, and asthma and related allergic disorders. A statement of the World Allergy Organization. World Allergy Organ J. 2015 Jul 14;8(1):25. doi: 10.1186/s40413-015-0073-0. eCollection 2015. PMID 26207160
- [Background] Li N, Georas S, Alexis N, Fritz P, Xia T, Williams MA, Horner E, Nel A. A work group report on ultrafine particles (American Academy of Allergy, Asthma & Immunology): Why ambient ultrafine and engineered nanoparticles should receive special attention for possible adverse health outcomes in human subjects. J Allergy Clin Immunol. 2016 Aug;138(2):386-96. doi: 10.1016/j.jaci.2016.02.023. Epub 2016 Apr 6. PMID 27130856
- [Background] Krishnan S, Panacherry S. Asthma, Environment and Pollution: Where the Rubber Hits the Road. Indian J Pediatr. 2018 Oct;85(10):893-898. doi: 10.1007/s12098-018-2691-3. Epub 2018 May 30. PMID 29845404
- [Background] Murrison LB, Brandt EB, Myers JB, Hershey GKK. Environmental exposures and mechanisms in allergy and asthma development. J Clin Invest. 2019 Apr 1;129(4):1504-1515. doi: 10.1172/JCI124612. Epub 2019 Feb 11. PMID 30741719
- [Background] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908